CLINICAL TRIAL: NCT06787469
Title: Clinical Performance of CAD/CAM Hard Hybrid Ceramic Overlays on Endodontically Treated Molars Using Bioactive Versus Conventional Self-Adhesive Resin Cement: Two-Year Randomized Clinical Trial
Brief Title: Comparison of the Clinical Performance of High Strength Hybrid Ceramic Indirect Restorations Cemented on Endodontically Treated Teeth Using Bioactive Versus Conventional Self Adhesive Resin Cements.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Nabil Hassan Shalaby, Assistant Lecturer - Conservative Dentistry Department - MIU, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANCU-8-1-2025
Record Dates: First submitted 2025-01-16; First posted 2025-01-22 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Endodontically Treated Molar
Keywords: Resin Cement; SHOFU; Bioactive Resin Cement; SPRG; S-PRG; Endodontically treated teeth; BeautiLink SA
MeSH Terms: conditions — Tooth, Nonvital | interventions — Resin Cements

STUDY DESIGN:
Intervention Model Description: This study will be conducted on the form of a randomized controlled, unicenter, clustered two-arm superiority trial with a 1:1 allocation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Indirect Restorations cemented using Coltene Solocem Resin Cement (Active Comparator)
  Interventions: Other: Resin Cement
- Indirect Restorations cemented using SHOFU BeautiLink Resin Cement (Active Comparator)
  Interventions: Other: Resin Cement

INTERVENTIONS:
Other: Resin Cement — Bioactive self adhesive resin cement (SHOFU BeautiLink) used to cement indirect restorations to endodontically treated molars.
  Arms: Indirect Restorations cemented using SHOFU BeautiLink Resin Cement
Other: Resin Cement — Self adhesive resin cement
  Arms: Indirect Restorations cemented using Coltene Solocem Resin Cement

SUMMARY:
Cementation of indirect restoration is a determinant of the success or failure of the fabricated restoration and consequentially the entire tooth. While there are numerous commercially available resin cements in the dental market, not all have been sufficiently assessed with significant follow up periods to clinically determine their success or failure. As such, this research will be conducted to elucidate if there is a viability to the cementation of indirect hybrid ceramic blocks over endodontically treated teeth using bioactive self-adhesive resin cement and determining whether it provides a clinical advantage and improved restoration serviceability in the oral cavity.

ELIGIBILITY:
Inclusion Criteria:

* Patient Related Criteria:
* Adult patients (age: 21-50 years) of both genders.
* Able to tolerate necessary restorative procedures.
* Willing to sign the informed consent.
* Accepts the follow-up period.

Tooth Related Criteria:

* Endodontically treated first and second permanent molars.
* Access cavities with one missing proximal wall i.e. Occluso-mesial/distal cavities
* Patients with proper oral hygiene

Exclusion Criteria:

* Endodontically treated anterior, premolar and third molar teeth
* Badly broken-down teeth
* Hopelessly carious/destructed teeth necessitating extraction
* Mobile teeth, indicating periodontal disease or trauma.
* External or internal resorption.
* Cervical carious lesions
* Medically compromised patients
* Patients with known allergies to Latex and/or resinous material

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-23 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Modified USPHS Criteria | 2 years

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR